CLINICAL TRIAL: NCT03008356
Title: L-Carnitine Supplementation With and Without Health Coaching for Fatigue in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: L-carnitine for Fatigue in COPD
Acronym: LC4COPD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-005732
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Copd; Fatigue
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fatigue | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- L-carnitine (Experimental): Oral L-carnitine 1000mg twice daily
  Interventions: Dietary Supplement: L-carnitine 1000 mg twice daily
- L-carnitine + health coaching (Experimental): Oral L-carnitine 1000mg twice daily and weekly 10-15 minute health coaching calls
  Interventions: Dietary Supplement: L-carnitine 1000 mg twice daily; Behavioral: Weekly health coaching calls
- Placebo (Placebo Comparator): Placebo capsules twice daily
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: L-carnitine 1000 mg twice daily — Oral L-carnitine to be taken twice daily for 8 weeks
  Arms: L-carnitine; L-carnitine + health coaching
Behavioral: Weekly health coaching calls — Weekly health coaching calls lasting 10-15 minutes
  Arms: L-carnitine + health coaching
Dietary Supplement: Placebo capsules
  Arms: Placebo

SUMMARY:
supplementation with L-carnitine that is available both as an FDA-approved therapy for primary carnitine deficiency, as well as widely available as an over-the-counter ergogenic aid will improve wellbeing and function measured by questionnaires in patient with chronic obstructive pulmonary disease (COPD).

based on our review of literature that addition of health coaching (HC) to L-carnitine will yield greater gains.

ELIGIBILITY:
Inclusion criteria:

- COPD patients with a positive screen for fatigue

Exclusion criteria:

* Vulnerable population - pregnant women, prisoners, unable to provide consent
* Pre-menopausal/breastfeeding women (pregnancy category B)
* Thyroid disease
* Anticoagulation therapy
* Decompensated cardiac disease
* Chronic Kidney Disease (CKD4 or above)
* Known seizure disorder
* Active malignancy
* Exacerbation of underlying pulmonary disease or acute illness in the 6 weeks before screening
* Enrollment in the past 6 weeks or currently in a cardiac or pulmonary rehab program or other physical fitness class(es).
* Difficulty with swallowing pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in Exercise Capacity as Measured by the Six Minute Walk Test (6MWT) | baseline, end of 8 week intervention
  The 6MWT is a widely studied, standardized and widely utilized test that evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. The self-paced 6MWT assesses the submaximal level of functional capacity. Most patients do not achieve maximal exercise capacity during the 6MWT; instead, they choose their own intensity of exercise and are allowed to stop and rest during the test.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life as Measured by the Chronic Respiratory Questionnaire (CRQ) | baseline, end of 8 week intervention
  The CRQ is a widely utilized and validated interviewer-administered questionnaire measuring both physical and emotional aspects of chronic respiratory disease. There are 20 questions, with each item graded on 7-point Likert scale. Scores can range from 20 to 100. Higher scores indicate better quality of life.
Change in Physical Fatigue as Measured by the Chalder Fatigue Questionnaire (CFQ-11) | baseline, end of 8 week intervention
  The CFQ-11 is a well-known, widely utilized and validated self-administered questionnaire for measuring the extent and severity of fatigue. The scoring incorporates two self-assessment scales measuring components indicative of physical fatigue [8 items] and mental fatigue [5 items]. The 11 individual items are scored from 0 (better than usual) to 3 (much worse than usual); total score range: 0-33.
Physical Activity as Measured by the SenseWear Armband | end of 8 week intervention
  The SenseWear Armband system (Temple Healthcare) is a versatile arm-band monitor allowing convenient and accurate collection of raw data regarding energy expenditure, sleep duration and quality, physical activity and movement in subjects in a free-living environment, allowing them to go about their normal daily activities. Patients will be shown how to wear the activity monitor and be asked to use it for at least 5 days for 23 hours a day. They will be provided instructions and pre-paid shipping materials for wear and return of the monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No